CLINICAL TRIAL: NCT03427957
Title: Evaluation of a New Hysteroscopic Grasper for Endometrial Biopsy in Post-menopausal Patients With Vaginal Bleeding and/or Endometrial Thickness
Brief Title: Evaluation of a New Hysteroscopic Grasper for Endometrial Biopsy in Post-menopausal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Antonio Simone Laganà, Medical Doctor, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HYGREB-1
Record Dates: First submitted 2018-01-19; First posted 2018-02-09 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Post-Menopausal Bleeding; Post-Menopausal Endometrial Thickness
Keywords: Hysteroscopy; Endometrial biopsy; Menopause

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Patients will be blinded to the type of grasper used to perform hysteroscopic endometrial biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- New hysteroscopic grasper (Experimental): Patients allocated in this group will undergo hysteroscopic endometrial biopsy through the new grasper with knurled terminal end and cutting jaws.
  Interventions: Diagnostic Test: Endometrial biopsy with the new hysteroscopic grasper with knurled terminal end and cutting jaws
- Classic spoon grasper (Active Comparator): Patients allocated in this group will undergo hysteroscopic endometrial biopsy through the classic spoon grasper.
  Interventions: Diagnostic Test: Endometrial biopsy with the hysteroscopic spoon grasper
- Classic alligator grasper (Active Comparator): Patients allocated in this group will undergo hysteroscopic endometrial biopsy through the classic alligator grasper.
  Interventions: Diagnostic Test: Endometrial biopsy with the hysteroscopic alligator grasper

INTERVENTIONS:
Diagnostic Test: Endometrial biopsy with the new hysteroscopic grasper with knurled terminal end and cutting jaws — Hysteroscopic endometrial biopsy performed through the new grasper with knurled terminal end and cutting jaws.
  Arms: New hysteroscopic grasper
Diagnostic Test: Endometrial biopsy with the hysteroscopic spoon grasper — Hysteroscopic endometrial biopsy performed through the spoon grasper.
  Arms: Classic spoon grasper
Diagnostic Test: Endometrial biopsy with the hysteroscopic alligator grasper — Hysteroscopic endometrial biopsy performed through the alligator grasper.
  Arms: Classic alligator grasper

SUMMARY:
Hysteroscopic endometrial biopsy is usually performed through the classic spoon grasper. Recently, a new hysteroscopic grasper with knurled terminal end and cutting jaws was designed, in order to improve feasibility of the procedure, reduce its duration and the discomfort for the patients.

This study aims to compare the outcomes of the three hysteroscopic graspers for endometrial biopsy in post-menopausal patients.

DETAILED DESCRIPTION:
Diagnostic hysteroscopy is currently the gold standard method to evaluate uterine cavity and tubal ostia, allowing also the visualization of vaginal walls and the cervical canal. Compared to the other available diagnostic techniques, hysteroscopy has the advantage of directly visualization the anatomical area to be investigated and allows to perform biopsy. The possibility of hysteroscopy-guided biopsy sampling is particularly important in order to get histological diagnosis. As recently suggested, the hysteroscopic biopsy of the endometrium has diagnostic accuracy of 90% for post-menopausal endometrial cancer.

Currently, most diagnostic hysteroscopies are performed in outpatient setting, without anesthesia, using modern hysteroscopes with a 1.67 mm working channel. In particular, endometrial biopsy is usually performed through the classic spoon grasper or alligator grasper. Recently, a new hysteroscopic grasper with knurled terminal end and cutting jaws was designed, in order to improve feasibility of the procedure, reduce its duration and the discomfort for the patients.

This study aims to compare the outcomes of the three hysteroscopic graspers for endometrial biopsy in post-menopausal patients.

ELIGIBILITY:
Inclusion Criteria:

* Physiologic menopause
* Vaginal bleeding or endometrial thickness (>5 mm)

Exclusion Criteria:

* Hormonal replacement therapies
* Other known causes of vaginal/cervical bleeding
* Suspected or known cancer(s)
* Premature or iatrogenic menopause
* Uterine cervix stenosis

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Duration of the hysteroscopy | During the hysteroscopy
  Duration of the hysteroscopic procedure, expressed in minutes and seconds.
Pain perceived by the patient | During the hysteroscopy
  Subjective evaluation of the pain perceived by the patient during the procedure, expressed through a 0-10 Visual Analogue Scale (VAS) score, where 0 means "No pain" and 10 "The worst imaginable pain".

SECONDARY OUTCOMES:
Number of attempts | During the hysteroscopy
  Number of attempts necessary to perform the biopsy
Size of the specimen | During the hysteroscopy
  Size of the specimen obtained through biopsy, expressed in mm2
Feasibility assessment by the operator | During the hysteroscopy
  Subjective assessment by the operator of the feasibility of performing the biopsy, expressed through a 0-10 Visual Analogue Scale (VAS) score, where 0 means "No feasible at all" and 10 "The most feasible event I could imagine".
Precision | During the hysteroscopy
  Subjective assessment by the operator of the precision of the biopsy, expressed through a 0-10 Visual Analogue Scale (VAS) score, where 0 means "No precise at all" and 10 "The most precise event I could imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Simone Laganà, M.D., Ph.D., Principal Investigator — Università degli Studi dell'Insubria; Salvatore Giovanni Vitale, M.D., Ph.D., Principal Investigator — University of Catania
Locations (2):
- Italy (2):
  - University of Catania, Catania
  - University of Insubria, Varese

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vitale SG, Lagana AS, Caruso S, Garzon S, Vecchio GM, La Rosa VL, Casarin J, Ghezzi F. Comparison of three biopsy forceps for hysteroscopic endometrial biopsy in postmenopausal patients (HYGREB-1): A multicenter, single-blind randomized clinical trial. Int J Gynaecol Obstet. 2021 Dec;155(3):425-432. doi: 10.1002/ijgo.13669. Epub 2021 Apr 4. PMID 33686708